CLINICAL TRIAL: NCT01624714
Title: Phase I Trial Monitoring Efficacy and Safety in Treatment of Alemtuzumab Naive Subjects and Data Collecting and Monitoring of Alemtuzumab Experienced Subjects With Refractory Multiple Sclerosis
Brief Title: Study of Alemtuzumab in Treatment Refractory MS Subjects/Alemtuzumab Naive & Alemtuzumab Experienced Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samuel Forrester Hunter, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Samuel Forrester Hunter, MD, PhD, President, Advanced Neurosciences Institute
Organization: Advanced Neurosciences Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPI-004
Record Dates: First submitted 2012-06-18; First posted 2012-06-21 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Sclerosis
Keywords: Treatment Refractory
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alemtuzumab Naive (Experimental): Alemtuzumab Subjects (30) with prior treatment refractoriness and treatment experience EDSS 3.0-7.0 inclusive, without contraindications to alemtuzumab
  Interventions: Drug: Alemtuzumab; Drug: Alemtuzumab immunotherapy
- Alemtuzumab Experienced (Experimental): Subjects with treatment refractory MS and prior alemtuzumab therapy (30)
  Interventions: Drug: Alemtuzumab; Drug: Alemtuzumab immunotherapy

INTERVENTIONS:
Drug: Alemtuzumab — alemtuzumab 12 mg IV x 5 daily doses at baseline, alemtuzumab 12 mg IV x 3 daily doses at month 12
  Other Names: Campath; Lemtrada
Drug: Alemtuzumab immunotherapy — Alemtuzumab 60 mg over 5 days for first annual cycle, then 36 mg over 3 days for subsequent annual cycle, and as needed cycles in subsequent years.

SUMMARY:
The purpose of this study is to treat prospectively documented clinic patients with treatment-refractory multiple sclerosis that are naïve to alemtuzumab. Alemtuzumab shows efficacy and rate of serious adverse events (SAEs) which is equivalent or better than standard of care treatment strategies used previously for treatment-refractory multiple sclerosis.

DETAILED DESCRIPTION:
Hypothesis Alemtuzumab manifests efficacy (e.g. improved MS Severity score, and treatment stability in relapse rate and Expanded Disability Status Scale [EDSS] progression) and serious adverse events (SAEs) equivalent or better than standard of care treatment strategies used prior to treatment for treatment-refractory multiple sclerosis.

Objectives Treat prospectively documented clinic patients treatment-refractory multiple sclerosis that are naïve to alemtuzumab.

Obtain retrospective disability, relapse, and adverse events in alemtuzumab-experienced subjects previously treated outside of clinical trial settings for treatment-refractory MS.

Obtain prospective safety and efficacy data for multiple sclerosis symptoms, disability, and adverse effects following the use of alemtuzumab for treatment-refractory MS in a population with exposures to prior cytotoxic and monoclonal antibody therapy.

Transition alemtuzumab-experienced clinic patients into a clinical trial setting for additional treatment with alemtuzumab as needed for refractory MS.

Coprimary outcomes will be: change in EDSS and converted EDSS to MS Severity scale.

Secondary outcomes: changes in annualized relapse rate, days of high dose corticosteroids, MRI-based cerebral volumes and burden of disease (in selected subjects), serious adverse events, and corticosteroid use. A questionnaire will be used to assess patient satisfaction with alemtuzumab as compared to prior therapies.

Safety outcomes will be assessed and tabulated.

ELIGIBILITY:
Inclusion Criteria:

* This trial treats subjects with relapsing variants of MS, including relapsing-remitting, progressive-relapsing, transitional, or secondary progressive MS, not amenable to other aggressive therapy, prior relapses, EDSS 2.5-7.0 inclusive. Most will have generally moderate to severe disability at EDSS >3 (EDSS 2.5-3 if significant cognitive complaints or MRI activity). Alemtuzumab experienced subjects at any EDSS level previously treated with alemtuzumab outside of a clinical trial are also eligible.

Inclusion Criteria for Alemtuzumab Experienced Subjects:

* All clinic patients who have been treated with alemtuzumab with our clinic method will be offered participation in the study, and may leave the study if desired after collection of data. Subjects wishing to sign informed consent but who have moved out of the region and are unable to be seen personally may be interviewed by telephone and included in the database after signing informed consent.

Exclusion Criteria:

* Subjects are excluded if they have purely slowly progressive or definite primary progressive MS (e.g. slowly progressive corticosteroid unresponsive myelopathy) with no documented recent relapses, advanced age (over 75 years), legal minor status, or a recognized contraindication to alemtuzumab (active infection, malignancy (other than considered surgical cures by oncologist or basal cell carcinoma), uncontrolled bleeding disorder, planned pregnancy in immediate future or unwillingness to use contraception, or if they are in another alemtuzumab clinical trial.
* Prior autoimmunity which is in remission or controlled will be considered at the investigator's discretion.
* Our clinic experience is that prior Grave's disease is not a contraindication to alemtuzumab therapy.
* We have not previously excluded patients from alemtuzumab on the basis of any humoral immune marker (e.g. anti-thyroid), and therefore do not plan to perform such testing in screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in Neurostatus Expanded Disability Status Scale | Baseline and every 6 months over 5 years
Change in MS Severity Scale | Baseline and every 6 months for 5 years

SECONDARY OUTCOMES:
Change in annualized relapse rate | Every 6 months during study
Number of treatment days with high dose corticosteroids | Every 6 months during study
Rate of serious adverse events | Duration of study
MRI-based cerebral volumes and burden of disease (in selected subjects) | Baseline and yearly X 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel F Hunter, MD, Principal Investigator — Advanced Neurosciences Institute (ANI)
Locations (1):
- Advanced Neurosciences Institute, Franklin, Tennessee, United States